CLINICAL TRIAL: NCT03740386
Title: Phentolamine Mesylate as a Reversal of Local Anesthesics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: León Formación (Other)
Responsible Party: Principal Investigator, alejandro gago garcia, Assintant professor, León Formación
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LeonFormacion
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia, Local
Keywords: phentolamine mesylate; reverse local anesthesia
MeSH Terms: interventions — Phentolamine

STUDY DESIGN:
Intervention Model Description: Three randomized groups
Who Masked: Participant, Investigator
Masking Description: We use a program to randomize three groups. Double blind study No sham or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lidocaine (Experimental): lidocaine 2% 1:80000
  Interventions: Drug: Phentolamine Mesylate 0.235 MG/ML [OraVerse]
- articaine (Experimental): articaine 4% 1:200000
  Interventions: Drug: Phentolamine Mesylate 0.235 MG/ML [OraVerse]
- bupivacaine (Experimental): bupivacaine 0,5% 1:200000
  Interventions: Drug: Phentolamine Mesylate 0.235 MG/ML [OraVerse]

INTERVENTIONS:
Drug: Phentolamine Mesylate 0.235 MG/ML [OraVerse] — compare effect of phentolamine mesylate in three arms

SUMMARY:
Oraverse © (Phentolamine mesylate) is a product designed to reverse the effect of local anesthetics used in dentistry. Its main objective is to reduce the postoperative period during which the patient suffers from the lack of sensitivity in the perioral soft tissues, it is an obvious discomfort, a difficulty to speak or eat, and sometimes a risk of self-injury in the lips and / or tongue .

The product was approved by the FDA in 2008 although the introduction in Spain has not occurred until December 2015. There are numerous studies that support its use, its effectiveness and safety, although none of the Spanish population, who have not yet had the opportunity to experience it.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY:

To analyze the response of Oraverse in patients receiving complete oral disinfection treatment, after administration of Lidocaine 2% 1/80000, Articaine 4% 1/200000 or Bupivacaine 0,5% 1:200000 in mandible, in comparison with the contralateral control side.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosticated to receive dental treatment according to Leonformacion's criteria

Exclusion Criteria:

* Hepatic or renal patient
* Fertility treatment, pregnancy or lactation
* Treatment with oral anticoagulants
* Patients with known allergies to anesthetics, excipients or phentolamine mesylate
* Patients with previous facial paresthesia
* Patients who had taken any painkiller or anti-inflammatory the day before
* Patients in which the anesthetic technique fails or has to be reinforced with more than two carpules

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
time lip recovery fron local anesthesia | 1 day
  self reported lip sensitivity by questionaire marking every 15 minutes

SECONDARY OUTCOMES:
Post intervention pain | 1 day
  visual analogue scale to measure pain: Line ranged from 1 to 10 units where 1 means no pain at all and 10 means the worst imaginable pain. Lower levels are good outcomes
post intervention bleeding | 1 day
  clinical assesment of post intervention bleeding when using phentolamine mesylate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Prados-Frutos JC, Rojo R, Gonzalez-Serrano J, Gonzalez-Serrano C, Sammartino G, Martinez-Gonzalez JM, Sanchez-Monescillo A. Phentolamine mesylate to reverse oral soft-tissue local anesthesia: A systematic review and meta-analysis. J Am Dent Assoc. 2015 Oct;146(10):751-9.e3. doi: 10.1016/j.adaj.2015.04.018. PMID 26409985
- [Result] Hersh EV, Moore PA, Papas AS, Goodson JM, Navalta LA, Rogy S, Rutherford B, Yagiela JA; Soft Tissue Anesthesia Recovery Group. Reversal of soft-tissue local anesthesia with phentolamine mesylate in adolescents and adults. J Am Dent Assoc. 2008 Aug;139(8):1080-93. doi: 10.14219/jada.archive.2008.0311. PMID 18682623
- [Result] Laviola M, McGavin SK, Freer GA, Plancich G, Woodbury SC, Marinkovich S, Morrison R, Reader A, Rutherford RB, Yagiela JA. Randomized study of phentolamine mesylate for reversal of local anesthesia. J Dent Res. 2008 Jul;87(7):635-9. doi: 10.1177/154405910808700717. PMID 18573982
- [Result] Fowler S, Nusstein J, Drum M, Reader A, Beck M. Reversal of soft-tissue anesthesia in asymptomatic endodontic patients: a preliminary, prospective, randomized, single-blind study. J Endod. 2011 Oct;37(10):1353-8. doi: 10.1016/j.joen.2011.06.019. Epub 2011 Aug 5. PMID 21924181
- [Result] Tavares M, Goodson JM, Studen-Pavlovich D, Yagiela JA, Navalta LA, Rogy S, Rutherford B, Gordon S, Papas AS; Soft Tissue Anesthesia Reversal Group. Reversal of soft-tissue local anesthesia with phentolamine mesylate in pediatric patients. J Am Dent Assoc. 2008 Aug;139(8):1095-104. doi: 10.14219/jada.archive.2008.0312. PMID 18682624
- [Result] Moore PA, Hersh EV, Papas AS, Goodson JM, Yagiela JA, Rutherford B, Rogy S, Navalta L. Pharmacokinetics of lidocaine with epinephrine following local anesthesia reversal with phentolamine mesylate. Anesth Prog. 2008 Summer;55(2):40-8. doi: 10.2344/0003-3006(2008)55[40:POLWEF]2.0.CO;2. PMID 18547152
- [Result] Hersh EV, Lindemeyer RG. Phentolamine mesylate for accelerating recovery from lip and tongue anesthesia. Dent Clin North Am. 2010 Oct;54(4):631-42. doi: 10.1016/j.cden.2010.06.004. PMID 20831927
- [Result] Elmore S, Nusstein J, Drum M, Reader A, Beck M, Fowler S. Reversal of pulpal and soft tissue anesthesia by using phentolamine: a prospective randomized, single-blind study. J Endod. 2013 Apr;39(4):429-34. doi: 10.1016/j.joen.2012.12.024. Epub 2013 Feb 11. PMID 23522530
- [Result] Daublander M, Liebaug F, Niedeggen G, Theobald K, Kurzinger ML. Effectiveness and safety of phentolamine mesylate in routine dental care. J Am Dent Assoc. 2017 Mar;148(3):149-156. doi: 10.1016/j.adaj.2016.11.017. Epub 2017 Jan 23. PMID 28126226